CLINICAL TRIAL: NCT03360864
Title: Impact of a Therapeutic Education Program in Patients With Non-radiological Spondyloarthritis Treated With Anti-tumor Necrosis Factor (TNF)
Brief Title: Influence of Therapeutic Education in Patients With Joint Inflammation Treated With a Biological Treatment
Acronym: ALSASP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6661
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Non-radiographic Spondyloarthritis
Keywords: Therapeutic education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Education Program (Experimental): Patient randomized in this arm will attend a 1 day long validated Therapeutic Education Program.
  This program will take place within 6 months after biologic treatment initiation.
  Interventions: Other: Education program
- No therapeutic Education Program (No Intervention): Patient randomized in this arm will not attend a Therapeutic Education Program within 12 months after biologic treatment initiation.

INTERVENTIONS:
Other: Education program — Patient will participate to a education program.
  Arms: Therapeutic Education Program

SUMMARY:
To describe, with a patient reported score (BIOSECURE), the influence of an approved therapeutic education program (TEP) in patients with joint inflammation requiring a biological treatment initiation.

The hypothesis is that patients attending the TEP will display better cognitive and adaptation competences than patients with no TEP.

Patient's reported quality of life, disease related stress management, treatment adherence, socio-demographic factors, biological home administration modalities and if the biologic treatment is maintained at 12 months, will also be described.

ELIGIBILITY:
Inclusion Criteria:

* Non-radiological spondyloarthritis diagnosis (ASAS criteria)
* Anti-TNFalpha biological treatment initiation required
* Adult patient (age>18years)
* Capacity to understand self-questionnaires and address questions
* Patient accepting to attend a therapeutic education program (TEP)

Exclusion Criteria:

* Previous Anti-TNFalpha biological treatment
* Previous attendance to a TEP concerning biological or spondyloarthritis
* Contraindication to Anti-TNFalpha treatment
* Associated and unbalanced diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-01-16 (Estimated); Study Completion 2023-01-16 (Estimated)

PRIMARY OUTCOMES:
BIOSECURE patient self-questionnaire | Change from Baseline Biosecure's score at 6 months and at 12 month after biological treatment initiation
  Patients will address questions and role play scenario evaluating cognitive and adaptive competences. The Biosecure score is between 0 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle SORDET, MD, Principal Investigator — CHU de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France